CLINICAL TRIAL: NCT00707564
Title: A Randomized, Self-Controlled Clinical Study of Hemostatic Efficacy of the HemCon Dental Dressing in a Population Treated With Anticoagulant Medications
Brief Title: Study of Hemostatic Efficacy of the HemCon Dental Dressing in a Population Treated With Anticoagulant Medications
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to enroll patient population
Sponsor: HemCon Medical Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-I-D-2
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Tooth Extractions
Keywords: hemostasis; tooth extractions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): HemCon Dental Dressing
  Interventions: Device: HemCon Dental Dressing
- 2 (Active Comparator): Gauze with pressure
  Interventions: Device: Gauze with pressure

INTERVENTIONS:
Device: HemCon Dental Dressing — The HemCon Dental Dressing is an oral wound dressing made of chitosan
  Other Names: HemCon Dental Dressing.
  Arms: 1
Device: Gauze with pressure — Gauze with pressure
  Other Names: Generic brand gauze with pressure.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if the HemCon Dental Dressing is effective in stopping bleeding during dental surgeries in patients taking anticoagulant medications.

DETAILED DESCRIPTION:
As the HemCon® Dental Dressing has been FDA cleared for use as a physical barrier for temporary protection of oral mucosal tissue and to provide pain relief, the proposed study will further investigate the safety and efficacy of hemostasis of the dressing for use in dental surgical procedures that do not require primary closure (suturing) such as tooth extractions. This protocol will specifically research the safety and efficacy of hemostasis within a population of subjects taking anticoagulant medications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are currently taking oral anticoagulant medications and eligible for surgery following standards of care
* Patients requiring a minimum of 2 tooth extraction procedures.
* Index pairing must reflect anatomically similar extraction locations
* 14 years of age or older
* Available for a minimum of one post operative evaluation approximately 7 days post surgery
* Extraction sites do not require primary closure or suturing
* Willingness and ability to provide informed consent/ assent

Exclusion Criteria:

* Scheduled to undergo a procedure other than tooth extractions
* In the Investigators opinion, dental surgery may pose a serious risk of uncontrollable bleeding due to anticoagulant use
* Scheduled to undergo 2 extractions, anatomically dissimilar
* Extraction procedures are expected to require primary closure or suture
* Unwilling or unable to provide informed consent/ assent
* Patients undergoing bisphosphonate therapy
* Patients not under current treatment with an oral anticoagulant medication
* Patients who have discontinued the use of anticoagulant medications for a minimum of 3 days prior to the planned surgical visit

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Time to hemostasis | minutes after application

SECONDARY OUTCOMES:
Incidence of post surgical sequela | 1 week post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jay Malmquist, DMD, Principal Investigator — Jay P. Malmquist, DMD, PC
Locations (2):
- United States (2):
  - Rodney Nichols, DMD, Milwaukie, Oregon
  - Jay P. Malmquist, DMD, Portland, Oregon